CLINICAL TRIAL: NCT00788528
Title: Open-Label Extension (OLE) Safety and Efficacy Study of Velneperit (S-2367) Following the Year-Long Controlled Clinical Trials of S-2367 in Obese Males and Females
Brief Title: Open-Label Extension (OLE) Study for Safety and Efficacy of Velneperit (S-2367) in Obese Subjects
Acronym: OLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0813A2825
Record Dates: First submitted 2008-11-07; First posted 2008-11-11 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental): 1600 mg S-2367 (velneperit)
  Interventions: Drug: S-2367 (velneperit)

INTERVENTIONS:
Drug: S-2367 (velneperit) — Tablet, 4 x 400 mg, taken once daily with morning meal, 54-weeks

SUMMARY:
The purpose of this open-label extension study is to evaluate the safety and efficacy of velneperit (S-2367) in obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Must have completed all randomized treatment visits in the reduced calorie diet (RCD, Shionogi protocol 0701A2823) or low calorie diet (LCD, Shionogi protocol 0702A2824) study up to and including Visit 13
* Medically stable throughout the controlled clinical trial treatment period and in otherwise good health, with no clinically significant findings from medical history, physical examination, 12-lead ECG, and vital signs
* Clinical laboratory evaluations (including clinical chemistry [fasted at least 8 hours], complete blood count, urinalysis, including creatine phosphokinase, amylase, lipase, lipid profile, insulin and Homeostatic Model Assessment of Insulin Sensitivity Index within the reference range for the test laboratory, unless deemed not clinically significant by the Investigator
* Males will be sterile or agree to continue to use an approved method of contraception. Some of the approved methods of contraception for males includes a surgically sterile (for at least 3 months prior to Visit 13/20) female sexual partner; a postmenopausal (for at least 1 year since last menstrual cycle) female sexual partner; a female sexual partner who uses (for at least previous 3 months prior to Visit 13/20 and during study) oral, implantable, transdermal, or injectable contraceptives; or use of the following double-barrier method: male condom with spermicide
* Females will be non-pregnant, non-lactating, and either postmenopausal for at least 1 year since last menstrual period, surgically sterile for at least 3 months prior to Visit 13/20, or agree to use an approved method of contraception. Some of the approved methods of contraception for females includes a sterile (for at least 3 months prior to Visit 13/20) male sexual partner; use of oral, implantable, transdermal, or injectable contraceptives; or use of one of the following double-barrier methods: intrauterine device with spermicide, diaphragm with spermicide, cervical cap with spermicide, female condom with spermicide, or a male condom with spermicide by the male sexual partner
* Able to understand and willing to sign an informed consent form and comply with all study procedures

Exclusion Criteria:

* History or clinical manifestations of significant metabolic, hepatic, immunological (e.g., human immunodeficiency virus/acquired immunodeficiency syndrome), renal, hematological, pulmonary, cardiovascular, gastrointestinal (GI), urological, neurological or psychiatric disorders
* Current abnormal ECG, which, in the Investigator's opinion, is clinically significant
* Current evidence of a psychological disorder, other than stable or controlled anxiety or depression including, but not limited to the schizophrenias. Treatment with an antidepressant or anxiolytic drug(s) will be permitted if the medication is not precluded / excluded by this protocol because of potential effects on body weight and is not expected to change during the remainder of this clinical protocol
* A score above 10 in either the Anxiety or Depression portions of the Hospital Anxiety and Depression Scale (HADS) at Visit 13/20. Subjects whose HADS score at Visit 13/20 exceeds 10 in either the Anxiety or Depression portions of the HADS will be allowed in the study only after they are examined and it is determined that the symptoms of anxiety and/or depression are not of a severity that is incompatible with further treatment with velneperit. Permission must also be obtained from the Sponsor or Sponsor's designated medical representative for subjects with scores above 10 on these HADS subscores
* Current obesity of endocrine origin
* Current Type 1 or Type 2 diabetes mellitus
* Current clinically significant hypertension, defined as blood pressure >160/90 mmHg for either the systolic or diastolic values in either the untreated or treated state
* Current or planned clinically significant GI surgery. Note: Appendectomy and cholecystectomy will be allowed
* Current or planned gastric bypass surgery, stomach banding surgery, or any other surgical procedure(s) that attempt to promote/aid weight loss. Note: Liposuction will be allowed if done more than 3 months prior to Study Visit 20
* Current polycystic ovarian syndrome
* Current or planned participation in any weight loss program outside of the program described in this open-label extension (OLE) study
* Current alcoholism or drug addiction/substance abuse. Note: Alcohol use during the study is allowed provided "routine" daily consumption is less than or equal to 2 units/day (1 unit is the equivalent of 12 oz. of beer, 5 oz. of wine, or 1.5 oz. of 80-proof distilled spirits [or equivalent]) and except that no alcohol consumption is allowed within 48 hours prior to blood collections for analysis of lipid profiles
* Current use of any tobacco-containing or nicotine-containing product (including cigarette, pipe, cigar, chewing, nicotine patch, or nicotine gum
* Current or planned participation in any other investigational study drug trial in which receipt of investigational study drug will occur
* Current or planned participation in any weight loss medication/product study in which receipt of weight loss medication/product will occur
* Current or planned use of any prescription or nonprescription over-the-counter (OTC) medication/product or herbal/phytotherapeutic/plant-derived medications/products that is intended to induce weight loss, appetite suppression, weight control or treat obesity, including, but not limited to, phentermine, sibutramine, orlistat, ephedra, rimonabant and other anorexogenics and/or stimulants, as well as topiramate, etc. Note: Use of any other medications/products for weight control, appetite suppression, treatment of obesity is prohibited during the course of this OLE study
* Current or planned use of chronic medications/products that are known to cause weight gain during the entire OLE study. The list includes but is not limited to amitriptyline (ELAVIL), paroxetine (PAXIL), setraline (ZOLOFT), and mirtazepine (REMERON). Additional clarification is provided in the concomitant medications section and Appendix B and updates or clarifications to these sections. Investigators are to discuss with the Sponsor's Medical Monitor any concomitant medications about which they are uncertain
* Current or planned use of any prescription or non-prescription OTC medications/product, unless deemed acceptable by the Investigator. Some examples of allowed medications are stable use (during RCD or LCD Study) of: hormone replacement therapy (e.g., for postmenopausal women); antihypertensive agents (e.g., for hypertensive subjects); statins (e.g., for hyperlipidemia); thyroid replacement therapy (e.g., for hypothyroid subjects and provided thyroid replacement therapy has been stable during the RCD or LCD study and no clinically significant changes in thyroid stimulating hormone and/or free thyroxine occur[s] during the study); oral, implantable, transdermal, or injectable contraceptive(s), etc. Anticholinergics (if used acutely), centrally acting antihistamines, and anti-inflammatories will also be allowed. Continued, stable, moderate use (during the RCD or LCD study) of vitamins and minerals is allowed and additional use of multivitamin-mineral supplements (non-herbal) may be allowed by the Investigator (or designee) as part of the study diet program
* Planned donation of blood or blood products during the entire OLE study
* Current poor peripheral venous access that would preclude blood collection
* Any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 766 (Actual)
Dates: Start 2008-08; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Efficacy assessment: The change in body weight over the 54-week active therapy phase of the study is the primary efficacy variable | 54 weeks
Treatment-emergent adverse events are summarized by system/organ class and preferred term using MedDRA. Safety assessments included clinical laboratory evaluations, vital signs, 12-lead electrocardiogram, physical examination, and reported adverse events | From the first dose of OLE study drug at Visit 20 until 30 days after the last dose of study drug

SECONDARY OUTCOMES:
Efficacy assessment: Secondary efficacy variables included analyses of body weight, body mass index, waist circumference, metabolic indexes, psychological variables, and dosage | Over the 54-week active therapy phase of the OLE study
Pharmacokinetic assessment: Pharmacokinetic trough levels were calculated based on the plasma concentrations. The data were analyzed at each interval and across intervals. Trough levels were correlated with dose, if appropriate | Weeks 3, 24, and 54

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (70):
- United States (70):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Hot Springs, Arkansas
  - Carmichael, California
  - Fountain Valley, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Stamford, Connecticut
  - Waterbury, Connecticut
  - Coral Gables, Florida
  - Jacksonville, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Stuart, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Gurnee, Illinois
  - Springfield, Illinois
  - Evansville, Indiana
  - Shawnee Mission, Kansas
  - Wichita, Kansas
  - Lexington, Kentucky
  - Boston, Massachusetts
  - Milford, Massachusetts
  - South Dartmouth, Massachusetts
  - Brooklyn Center, Minnesota
  - Gulfport, Mississippi
  - Kansas City, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Berlin, New Jersey
  - Edison, New Jersey
  - Endwell, New York
  - Manlius, New York
  - Rochester, New York
  - Burlington, North Carolina
  - Concord, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Mogadore, Ohio
  - Yukon, Oklahoma
  - Bensalem, Pennsylvania
  - Cranston, Rhode Island
  - Greenville, South Carolina
  - Mt. Pleasant, South Carolina
  - Bristol, Tennessee
  - Burns, Tennessee
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Houston, Texas
  - Jackson, Texas
  - New Braunfels, Texas
  - San Antonio, Texas
  - West Jordan, Utah
  - Richmond, Virginia
  - Renton, Washington
  - Green Bay, Wisconsin
  - Wauwatosa, Wisconsin